CLINICAL TRIAL: NCT06535347
Title: Nudging High-acuity Emergency Department Patients to Schedule a Follow-up Visit With a Primary Care Provider or Specialist Following Discharge to Decrease Emergency Department Utilization
Brief Title: Nudging High-acuity Emergency Department Patients to Schedule a Follow-up Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, ‪Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0412
Record Dates: First submitted 2024-07-08; First posted 2024-08-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Emergency Service, Hospital
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Masking Description: Patients will be aware of their own messages but will not be aware of other messages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): This arm will receive no intervention outside of usual care.
- Experimental: Schedule Follow-Up Visit - 1 message (Experimental): This arm will receive a text message (at 1 day post-ED discharge) and information added to the patient's after visit summary providing a number and patient portal hyperlink via which to schedule an ED follow-up appointment.
  Interventions: Behavioral: Information about scheduling a follow-up appointment
- Experimental: Schedule Follow-Up Visit - 2 messages (Experimental): This arm will receive text messages (at 1 day and 8 days post-ED discharge) and information added to the patient's after visit summary providing a number and patient portal hyperlink via which to schedule an ED follow-up appointment.
  Interventions: Behavioral: Information about scheduling a follow-up appointment

INTERVENTIONS:
Behavioral: Information about scheduling a follow-up appointment — Text message(s) will be sent following discharge from the emergency department, along with an after visit summary.
  Other Names: Text messages; Information
  Arms: Experimental: Schedule Follow-Up Visit - 1 message; Experimental: Schedule Follow-Up Visit - 2 messages

SUMMARY:
The goal of this campaign is to reduce unnecessary emergency department (ED) visits by encouraging patients with high acuity visits to follow up with an appropriate primary care provider (PCP) or specialist and therefore obtain appropriate care outside of the ED. In this campaign, patients will be assigned to receive or not receive outreach following ED discharge that is aligned with the goal. Outreach will occur via a text message and information added to the patient's after visit summary, and will include a contact number to schedule and hyperlink to allow self-scheduling. The study will assess whether ED use differs across patients in different outreach conditions. It will also examine whether patients followed through on the calls to action in the messages differently across conditions.

DETAILED DESCRIPTION:
Enrollment will conclude when either 7500 participants have been enrolled or after 120 days, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* ED visit rated as high acuity (level L2 or L3)
* Discharged from ED in past 24 hours
* Attributed to a Geisinger PCP in Community Medicine Service Line

Exclusion Criteria:

* Have an appointment scheduled within 7 days following discharge with a primary care provider or specialist
* Institutionalized
* Cannot be contacted via the communication modality being used in the study (i.e., SMS), due to insufficient/missing contact information in the electronic health record or because the patient opted out
* Admitted to hospital
* Eloped from ED
* Left ED without being seen
* Deceased prior to messaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6814 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-04-06 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Return to ED | within 120 days following day of discharge
  ED visit (yes/no)

OTHER OUTCOMES:
PCP/specialist appointment made | within 7 days following day of discharge
  PCP or specialist appointment made
PCP/specialist appointment made | within 14 days following day of discharge
  PCP or specialist appointment made
PCP/specialist appointment made | within 30 days following day of discharge
  PCP or specialist appointment made
PCP/specialist appointment made | within 60 days following day of discharge
  PCP or specialist appointment made
PCP/specialist appointment attended | within 7 days following day of discharge
  PCP or specialist appointment attended
PCP/specialist appointment attended | within 14 days following day of discharge
  PCP or specialist appointment attended
PCP/specialist appointment attended | within 30 days following day of discharge
  PCP or specialist appointment attended
PCP/specialist appointment attended | within 60 days following day of discharge
  PCP or specialist appointment attended

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT06535347/Prot_SAP_000.pdf